CLINICAL TRIAL: NCT03773354
Title: Somatic Symptom and Related Disorders: A Pilot Treatment Group and Mixed-Methods Investigation
Brief Title: Somatic Symptom and Related Disorders: A Treatment Group and Mixed-Methods Investigation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Emily MacKillop, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5498
Record Dates: First submitted 2018-12-05; First posted 2018-12-12 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Somatic Symptom Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): There is no control group for this study, and all participants receive the intervention. Although a few participants will be asked to give additional information during the intake and after the study concludes for quality improvement purposes. Effects of these additional interview questions will be considered during analysis
  Interventions: Behavioral: Cognitive-behavioural therapy group for individuals with somatic symptom disorders

INTERVENTIONS:
Behavioral: Cognitive-behavioural therapy group for individuals with somatic symptom disorders — The intervention is a cognitive-behavioural therapy group for designed for individuals with a formal diagnosis of a somatic symptom disorder (i.e., Somatic Symptom and Related Disorders from the DSM-5) who are interested in learning self-management skills to cope with somatic symptoms and reduce emotional dysregulation, increasing their understanding of factors that contribute to somatic symptoms, and learning relaxation skills to help reduce stress.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a new cognitive behavioural therapy (CBT) group for individuals with a somatic symptom disorder (i.e., Somatic Symptom and Related Disorders from the DSM-5). Patients with somatic symptom and related disorders are underserved by the medical system. Further, there is currently a paucity of research aimed at evaluating treatments for patients with somatic symptom disorders. The limited existing research literature supports CBT as an efficacious treatment in this population, but a standardized means of modifying CBT for somatic symptom disorders has not been developed, and it is unclear if group CBT is effective. In this study, the investigators will evaluate the effectives of a new six session CBT group designed specifically to address commonly-reported difficulties among individuals with somatic symptom disorders, such as somatic symptoms, psychological distress, and related cognitive interference. This study will allow us to validate a new intervention for somatic symptom disorders, and will help to fill the current void of evidence-supported evaluation and treatment protocols to better serve patients with somatic symptom disorders.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older,
2. formally diagnosed with a somatic symptom or related disorder,
3. registered patients of St. Joseph's Healthcare Hamilton, and
4. subjective psychological complaints and somatic complaints causing distress and/or functional impairment.

Exclusion Criteria: individuals with

1. acute and severe depression/suicidal ideation,
2. severe PTSD symptoms,
3. current psychosis,
4. current substance use disorder, or
5. severe cognitive impairment will be excluded from the study and referred to a more appropriate intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2019-12-03 (Estimated); Study Completion 2020-02-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline self-reported distress related to somatic symptoms at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Patient Health Questionnaire 15-Item (PHQ-15) Somatic Symptom Severity. Scores are added to form a total score ranging from 0-30 with higher values indicating more severe distress related to somatic symptoms.

SECONDARY OUTCOMES:
Baseline estimated level of intellectual ability | Week 1 (prior to intervention)
  Will be measured with the Advanced Clinical Solutions - Test of Premorbid Functioning (copyrighted), which results in a total raw score ranging from 0-70, and is normatively scored based on respondents' age resulting in standard scores (mean = 100). Higher values indicate a higher premorbid level of intellect.
Change from baseline intellectual functioning at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Wechsler Abbreviated Scale of Intelligence - 2nd Edition (copyrighted), which results in a total raw score (full scale intellectual quotient) ranging from 0-205, and is normatively scored based on respondents' age resulting in standard scores (mean = 100). Higher values indicate a higher level of intellect.
Baseline performance validity | Week 1 (prior to intervention)
  Measured with the Victoria Symptom Validity Test (copyrighted), which has two subtests of Easy Items (raw scores ranging from 0-24) and Hard Items (raw scores ranging from 0-24), which higher scores indicating better performance.
Performance validity at 6 weeks | Week 6 (post-intervention)
  Measured with the Victoria Symptom Validity Test (copyrighted), which has two subtests of Easy Items (raw scores ranging from 0-24) and Hard Items (raw scores ranging from 0-24), which higher scores indicating better performance.
Change from baseline auditory working memory at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Measured with the Digit Span subtest of the Wechsler Adult Intelligence Scale - 4th Edition (copyrighted), which results in three subtests (Digit Span Forward, Digit Span Backward, and Digit Span Sequencing), each ranging from a raw score of 0-16 and scored normatively resulting in scaled score (mean = 10). Higher scores indicate better performance.
Change from baseline visual attention and speed at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with Trails A & B. The participants' response time on each of the two tasks is scored normatively resulting in a t-score (mean = 50). Higher t-scores indicate better performance.
Change from baseline motor speed at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured on Grooved Pegboard. The time taken to complete the task with each hand will be normatively scored, resulting in a t-score. Higher t-scores are indicative of better performance.
Change from baseline verbal fluency at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with phonemic fluency (FAS) and semantic fluency (animals) tasks. The number of words they provide is normatively scored resulting in t-scores. Higher t-scores are indicative of better performance.
Change from baseline overall neurocognitive performance at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Repeatable Battery for the Assessment of Neuropsychological Status Update (copyrighted), which results in 12 subtests that are normatively scored, summed together, and normatively scored to result in a index score (mean = 100) with higher values indicating better performance.

OTHER OUTCOMES:
Baseline personality traits | Week 1 (prior to intervention)
  Will be measured with the Personality Assessment Inventory (copyrighted), which is a 344 item with 22 scales. Each question is answered on a 4-point Likert scale. Higher scores generally are indicative of greater symptom severity.
Change from baseline alcohol consumption at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Alcohol Use Disorders Identification Test (AUDIT), which is a 10-item questionnaire with a 5 point Likert scale. Questions are summed resulting in a total score ranging from 0-40, which higher numbers indicating greater alcohol consumption.
Change from baseline cannabis consumption at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Cannabis Use Disorders Identification Test - Revised (CUDIT-R), which is an 8-item questionnaire with a 5 point Likert scale. Questions are summed resulting in a total score ranging from 0-32, which higher numbers indicating greater cannabis consumption.
Change from baseline drug use at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Drug Use Disorders Identification Test (DUDIT), which is an 11-item questionnaire with a 5 point Likert scale. Questions are summed resulting in a total score ranging from 0-44, which higher numbers indicating greater drug use.
Change from baseline nicotine dependence at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with adapted version of the Fagerstrom Test for Nicotine Dependence (FTND), which is a 3-item questionnaire. Participants are asked open-ended questions regarding their quantity of cigarette consumption. Then they rank their willingness to cut down on a scale from 1-10, which 10 indicated highest readiness for change.
Change from baseline substance use at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with Nida Substance Use Checklist, which is a 5-point Likert scale with 6 items. Items are summed resulting in a total score ranging from 0-24, with higher scores indicating greater substance use.
Change from baseline readiness for change at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Readiness Ruler, which consists of 8 items rated on a 10 point Likert Scale. Items are summed and total scores range from 8-80, and higher scores indicate greater readiness for change.
Change from baseline problem gambling at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Problem Gambling Severity Index (PGSI), which consists of 9 items rated on a 4-point Likert Scale. Items are summed and total scores range from 0-27, with higher scores indicating more severe problem gambling.
Change from baseline symptoms of attention deficit/hyperactivity disorder at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Adult ADHD Self-Report Scale (ASRS-v1.1), which consists of 6 items rated on a 5 point Likert scale. Items are summed into a total score ranging from 0-24, with higher scores indicating more severe symptoms of ADHD.
Change from baseline depressive symptoms at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Patient Health Questionnaire - Depression (PHQ-D), which consists of 9 items rated on a 4 point Likert scale. Items are summed into a total score ranging from 0-27, with higher scores indicating more severe symptoms of depression.
Change from baseline symptoms of anxiety at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Generalized Anxiety Disorder 7-Item (GAD-7), which consists of 7 items rated on a 4 point Likert scale. Items are summed into a total score ranging from 0-21, with higher scores indicating more severe symptoms of anxiety.
Change from baseline symptoms of disordered eating at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Patient Health Questionnaire - Eating Disorders (PHQ - ED), which consists of 8 yes/no questions. Item endorsement is indicative of symptoms of disordered eating, and different items correspond with different eating disorders.
Change from baseline traits of borderline personality disorder at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the McClean Screening Instrument for Borderline Personality Disorder (MSI-BPD), which consists of 10 yes/no questions. The number of "yes" responses is added resulting in a total score ranging from 0-10, with higher scores indicating more features of borderline personality disorder.
Change from baseline prodromal symptoms at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Prodromal Questionnaire, which is a 16 item true/false questionnaire. The number of symptom endorsements are added resulting in a total score ranging from 0-16, with higher scores indicating more severe prodromal symptoms.
Change from baseline traumatic experiences at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Brief Trauma Questionnaire, which is a 10-item yes/no questionnaire. Items are summed to form a total score ranging from 0-10, with higher scores consistent with more traumatic event exposure.
Change from baseline post-traumatic stress disorder (PTSD) symptoms at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the PTSD Checklist for DSM-5 (PCL-5), which consists of 20 items rated on a 5 point Likert scale. The items are added resulting in a total score ranging from 0-80, with higher scores indicating more severe symptoms of PTSD.
Change from baseline indicators of traumatic brain injury at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Ohio State University Traumatic Brain Injury Identification Method (OSU-TBI), which consists of 5 yes/no questions. "Yes" responses are counted resulting in a total score from (0-5), with higher numbers indicating more indicators of traumatic brain injury.
Change from baseline perceived stress at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Perceived Stress Scale 4, which consists of 4 items rated on a 5 point Likert scale. Items are summed resulting in a total score ranging from 0-16, with higher scores indicating more perceived stress.
Change from baseline delay discounting ability at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the 5-Trial Adjusting Delay Discounting Task, in which participants are presented with five choice between hypothetical smaller-immediate and larger-delayed monetary rewards. Responses are summed resulting in a total score ranging from 1 hour to 25 years, and longer periods of time are indicative of greater delay discounting.
Change from baseline distress tolerance at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Distress Tolerance Scale - Shortened Version, which consists of 5 items rated on a 5 point Likert scale. Items are summed resulting in a total score ranging from 5-15 with higher scores corresponding to greater levels of distress tolerance.
Change from baseline impulsive behaviour at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Short Urgency, Premeditation (lack of), Perseverance (lack of), Sensation Seeking, Positive Urgency (UPPS-P) Impulsive Behaviour Scale, which consists of 20 items rated on a 4 point Likert scale. Items are summed together resulting in a total score ranging from 20-80, with higher values indicating more impulsive behaviour.
Change from baseline mindfulness at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Mindfulness Awareness Attention Scale (MAAS) - shortened version, which consists of 5 items rated on a 6 point Likert scale. Items are averaged resulting in a total score ranging from 1-6, with higher scores reflecting higher levels of dispositional mindfulness.
Change from baseline somatic symptom severity at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Patient Health Questionnaire 15-item Somatic Symptom Severity Scale, which consists of 15 items rated on a 3 point Likert scale. Items are added resulting in a total score ranging from 0-30, with higher score reflecting greater somatic symptom severity.
Change from baseline level of disability at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the World Health Organization Disability Assessment Schedule, which consists of 12 items rated on a 5 point Likert scale. Items are summed to form a total score ranging from 0-48, with higher scores reflecting a greater level of disability.
Change from baseline pain disability at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Pain Disability Index, which consists of 7 items rated on a 10 point Likert scale. Items are summed resulting in a total score ranging from 0-70, with higher scores indicating more pain disability.
Change from baseline pain self-efficacy at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Pain Self-Efficacy Questionnaire, which consists of 10 items rated on a 7 point Likert scale. Items are summed resulting in a total score ranging from 0-60, with higher scores reflecting greater pain self-efficacy.
Change from baseline resilience at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Brief Resilience Scale, which consists of 6 items rated on a 5 point Likert scale. Items are added forming a total score ranging from 0-24, which higher scores reflecting higher levels of resilience.
Change from baseline illness perception at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Illness Perception Questionnaire. First, participants are presented with 14 symptoms and asked to select whether or not they experience them (yes/no). Next, participants answer 38 questions regarding their illness perception on a 5 point Likert scale. Items on this subscale are summed (13 are reverse scored) resulting in total scores ranging from 0-152, with higher scores reflecting positive beliefs about the controllability of the illness and a personal understanding of the condition. Last, participants rate factors they believe to have contributed to their illness on a 5 point Likert scale.
Change from baseline recent life events at 6 weeks | Week 1 (prior to intervention), week 6 (post-intervention)
  Will be measured with the Schedule of Recent Events. Participants indicate how many times they experienced 42 potential life events within the preceding year. The frequency of each item is multiplied by the mean value provided and then scores are summed together. Higher scores are indicative of many recent stressful life events.

IPD SHARING:
Plan to Share IPD: No